CLINICAL TRIAL: NCT07100080
Title: IZABRIGHT-Lung01: A Randomized, Open-label, Phase 2/3 Study of Izalontamab Brengitecan (BMS-986507) Versus Platinum-based Chemotherapy in Patients With EGFR-mutated Non-small Cell Lung Cancer and Disease Progression on EGFR Tyrosine Kinase Inhibitor Therapy
Brief Title: Study of Izalontamab Brengitecan (BMS-986507) Versus Platinum-Pemetrexed for EGFR-mutated Non-small Cell Lung Cancer After Failure of EGFR TKI Therapy (IZABRIGHT-Lung01)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA244-0010; EU CTR (Other: 2025-521908-22); WHO (Other: U1111-1321-3429); CA2440010 (Other: Bristol-Myers Squibb Protocol ID)
Record Dates: First submitted 2025-07-31; First posted 2025-08-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Epidermal Growth Factor Receptor; Tyrosine Kinase Inhibitors; Osimertinib; Standard of Care; Lung Neoplasms; Antineoplastic Agents; Izalontamab brengitecan; Iza-bren; BL-B01D1; Carboplatin; Cisplatin; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Carboplatin; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Experimental)
  Interventions: Drug: Iza-bren
- Arm B (Experimental)
  Interventions: Drug: Iza-bren
- Arm C (Active Comparator)
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed
- Arm D (Experimental)
  Interventions: Drug: Iza-bren
- Arm E (Active Comparator)
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Iza-bren — Specified dose on specified days
  Other Names: BMS-986507; BL-B01D1; Izalontamab brengitecan
  Arms: Arm A; Arm B; Arm D
Drug: Carboplatin — Specified dose on specified days
  Arms: Arm C; Arm E
Drug: Cisplatin — Specified dose on specified days
  Arms: Arm C; Arm E
Drug: Pemetrexed — Specified dose on specified days
  Arms: Arm C; Arm E

SUMMARY:
A Study of Izalontamab Brengitecan (BMS-986507) versus Platinum-Pemetrexed for EGFR-mutated Non-small Cell Lung Cancer after failure of EGFR TKI Therapy

ELIGIBILITY:
Inclusion Criteria:

* Non-squamous NSCLC, not amenable to treatment in curative intent.
* Documented evidence of EGFR mutation (exon 19 deletion, L858R mutation).
* Progressive disease on a 3rd-generation (such as osimertinib, furmonertinib, lazertinib,...) EGFR-TKI-based mono- or combination therapy regimen as the most recent line of therapy in an adjuvant, locally advanced, or metastatic treatment setting.
* Eligible to receive a platinum-based doublet chemotherapy regimen (either cisplatin or carboplatin in combination with pemetrexed).

Exclusion criteria:

* Inadequate organ function and/or bone marrow reserve.
* Leptomeningeal metastases or spinal cord compression.
* Poorly controlled systemic medical conditions.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2031-05-15 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 3 Dose (RP3D) of BMS-986507 | Approximately 3 months after the first dose
  Phase 2
Progression-Free Survival (PFS) Assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) per blinded independent central review (BICR) | Up to 3 years
  Phase 3

SECONDARY OUTCOMES:
Objective Response (OR) Assessed by RECIST v1.1 per BICR | Up to 3 years
  Phase 2
PFS Assessed by RECIST v1.1 per BICR | Up to 3 years
  Phase 2
Overall Survival (OS) | Up to 5 years
  Phase 3
PFS Assessed by RECIST v1.1 per investigator assessment | Up to 3 years
  Phase 3
OR Assessed by RECIST v1.1 per BICR | Up to 3 years
  Phase 3
Disease Control Rate (DCR) Assessed by RECIST v1.1 per BICR | Up to 3 years
  Phase 3
Duration of Response (DOR) Assessed by RECIST v1.1 per BICR | Up to 3 years
  Phase 3
Time To Response (TTR) Assessed by RECIST v1.1 per BICR | Up to 3 years
  Phase 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (185):
- United States (27):
  - Local Institution - 0279, Irvine, California
  - Local Institution - 0154, Orange, California
  - Shaw Cancer Center, Edwards, Colorado
  - Local Institution - 0085, Gainesville, Florida
  - Local Institution - 0270, Atlanta, Georgia
  - Local Institution - 0143, Columbus, Georgia
  - Local Institution - 0153, Chicago, Illinois
  - Local Institution - 0282, South Portland, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Local Institution - 0276, Reno, Nevada
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Health, New York, New York
  - Local Institution - 0158, New York, New York
  - Local Institution - 0186, Rochester, New York
  - Local Institution - 0087, Cleveland, Ohio
  - Local Institution - 0038, Portland, Oregon
  - Local Institution - 0275, Portland, Oregon
  - Local Institution - 0171, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Local Institution - 0088, Pittsburgh, Pennsylvania
  - Local Institution - 0268, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Local Institution - 0025, Houston, Texas
  - Local Institution - 0173, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Local Institution - 0138, Richmond, Virginia
- Argentina (3):
  - Local Institution - 0008, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0004, ABB, Buenos Aires F.D.
  - Local Institution - 0094, Córdoba, Córdoba Province
- Belgium (5):
  - Local Institution - 0280, Wilrijk, Antwerpen
  - Local Institution - 0161, Auderghem, Bruxelles-Capitale, Région de
  - Local Institution - 0022, Yvoir, Namur
  - Local Institution - 0023, Ghent, Oost-Vlaanderen
  - Local Institution - 0024, Sint-Niklaas, Oost-Vlaanderen
- Canada (4):
  - Local Institution - 0190, Calgary, Alberta
  - Local Institution - 0183, Toronto, Ontario
  - Local Institution - 0184, Chicoutimi, Quebec
  - Local Institution - 0185, Montreal, Quebec
- Chile (3):
  - Local Institution - 0006, Santiago, Santiago Metropolitan
  - Local Institution - 0005, Santiago, Santiago Metropolitan
  - Local Institution - 0007, Santiago, Santiago Metropolitan
- China (20):
  - Local Institution - 0244, Beijing, Beijing Municipality
  - Local Institution - 0259, Chongqing, Chongqing Municipality
  - Local Institution - 0253, Fuzhou, Fujian
  - Local Institution - 0245, Jiangmen, Guangdong
  - Local Institution - 0271, Anyang, Henan
  - Local Institution - 0261, Luoyang, Henan
  - Local Institution - 0267, Jingzhou, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Local Institution - 0255, Changsha, Hunan
  - Local Institution - 0256, Xuzhou, Jiangsu
  - Local Institution - 0247, Nanchang, Jiangxi
  - Local Institution - 0246, Changchun, Jilin
  - Local Institution - 0257, Shenyang, Liaoning
  - Local Institution - 0248, Jinan, Shandong
  - Local Institution - 0250, Shanghai, Shanghai Municipality
  - Local Institution - 0258, Taiyuan, Shanxi
  - Local Institution - 0252, Hangzhou, Zhejiang
  - Local Institution - 0251, Linhai, Zhejiang
  - Local Institution - 0260, Nanning
  - Local Institution - 0249, Shanghai
- Colombia (4):
  - Local Institution - 0229, Valledupar, Cesar Department
  - Local Institution - 0228, Bogotá, Cundinamarca
  - Local Institution - 0227, Montería, Departamento de Córdoba
  - Local Institution - 0226, Cali, Valle del Cauca Department
- France (11):
  - Local Institution - 0014, Strasbourg, Alsace
  - Local Institution - 0017, Toulouse, Haute-Garonne
  - Local Institution - 0010, Lille, Hauts-de-France
  - Local Institution - 0018, La Tronche, Isère
  - Local Institution - 0170, Saint-Herblain, Loire-Atlantique
  - Local Institution - 0162, Bron, Rhône
  - Local Institution - 0019, Villejuif, Val-de-Marne
  - Local Institution - 0012, Marseille
  - Local Institution - 0278, Nantes
  - Local Institution - 0011, Paris
  - Local Institution - 0015, Paris
- Germany (14):
  - Local Institution - 0207, Esslingen am Neckar, Baden-Wurttemberg
  - Local Institution - 0238, Esslingen am Neckar, Baden-Wurttemberg
  - Local Institution - 0212, Stuttgart, Baden-Wurttemberg
  - Local Institution - 0236, Donauwörth, Bavaria
  - Local Institution - 0209, Oldenburg, Lower Saxony
  - Local Institution - 0213, Cologne, North Rhine-Westphalia
  - Local Institution - 0208, Chemnitz, Saxony
  - Local Institution - 0274, Kiel, Schleswig-Holstein
  - Local Institution - 0211, Berlin
  - Local Institution - 0215, Gauting
  - Local Institution - 0242, Hamburg
  - Local Institution - 0210, Heidelberg
  - Local Institution - 0239, Kassel
  - Local Institution - 0241, Ulm
- Greece (4):
  - Local Institution - 0054, Athens, Attikí
  - Local Institution - 0060, Chaïdári, Attikí
  - Local Institution - 0056, Thessaloniki, Kentrikí Makedonía
  - Local Institution - 0062, Thessaloniki, Thessaloníki
- India (9):
  - Local Institution - 0083, Ahmedabad, Gujarat
  - Local Institution - 0073, Ahmedabad, Gujarat
  - Local Institution - 0072, Gurugram, Haryana
  - Local Institution - 0069, Bengaluru, Karnataka
  - Local Institution - 0077, Mumbai, Maharashtra
  - Local Institution - 0071, Mumbai, Maharashtra
  - Local Institution - 0097, Nagpur, Maharashtra
  - Local Institution - 0070, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0078, Howrah, West Bengal
- Italy (8):
  - Local Institution - 0028, Ravenna, Emilia-Romagna
  - Local Institution - 0036, Aviano, Friuli Venezia Giulia
  - Local Institution - 0031, Orbassano, Piedmont
  - Local Institution - 0277, Candiolo, Torino
  - Local Institution - 0137, Avellino
  - Local Institution - 0032, Milan
  - Local Institution - 0034, Napoli
  - Local Institution - 0029, Parma
- Japan (15):
  - Local Institution - 0196, Nagoya, Aichi-ken
  - Local Institution - 0191, Kashiwa, Chiba
  - Local Institution - 0203, Tōon, Ehime
  - Local Institution - 0201, Kurume, Fukuoka
  - Local Institution - 0217, Sapporo, Hokkaido
  - Local Institution - 0199, Nishinomiya, Hyōgo
  - Local Institution - 0193, Yokohama, Kanagawa
  - Local Institution - 0192, Sendai, Miyagi
  - Local Institution - 0200, Kurashiki, Okayama-ken
  - Local Institution - 0198, Hirakata, Osaka
  - Local Institution - 0204, Ōsaka-sayama, Osaka
  - Local Institution - 0194, Ina-machi, Saitama
  - Local Institution - 0197, Hamamatsu, Shizuoka
  - Local Institution - 0195, Nagaizumi-cho,Sunto-gun, Shizuoka
  - Local Institution - 0202, Koto-ku, Tokyo
- Mexico (4):
  - Local Institution - 0225, Mexico City, Mexico City
  - Local Institution - 0224, Oaxaca City, Oaxaca
  - Local Institution - 0222, Chihuahua City
  - Local Institution - 0223, Mexico City
- Netherlands (3):
  - Local Institution - 0163, Harderwijk, Gelderland
  - Local Institution - 0216, Amsterdam, North Holland
  - Local Institution - 0164, Amsterdam, North Holland
- Norway (3):
  - Local Institution - 0103, Drammen, Buskerud
  - Local Institution - 0106, Bergen, Hordaland
  - Local Institution - 0105, Oslo
- Poland (3):
  - Local Institution - 0220, Lublin, Lublin Voivodeship
  - Local Institution - 0231, Gdynia, Pomeranian Voivodeship
  - Local Institution - 0219, Bydgoszcz
- Romania (8):
  - Local Institution - 0120, Bucharest, București
  - Local Institution - 0123, Bucharest, București
  - Local Institution - 0132, Florești, Cluj
  - Local Institution - 0130, Craiova, Dolj
  - Local Institution - 0115, Bucharest
  - Local Institution - 0133, Cluj-Napoca
  - Local Institution - 0124, Iași
  - Local Institution - 0119, Iași
- Singapore (2):
  - Local Institution - 0263, Singapore
  - Local Institution - 0262, Singapore
- South Korea (8):
  - Local Institution - 0089, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Local Institution - 0043, Goyang-si, Kyǒnggi-do
  - Local Institution - 0044, Seongnam, Kyǒnggi-do
  - Local Institution - 0046, Suwon, Kyǒnggi-do
  - Local Institution - 0095, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0045, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0092, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0042, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (10):
  - Local Institution - 0218, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0177, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0175, Madrid, Madrid, Comunidad de
  - Local Institution - 0206, Madrid, Madrid, Comunidad de
  - Local Institution - 0176, Madrid, Madrid, Comunidad de
  - Local Institution - 0181, Majadahonda, Madrid, Comunidad de
  - Local Institution - 0178, Málaga
  - Local Institution - 0182, Seville
  - Local Institution - 0180, Valencia
  - Local Institution - 0179, Zaragoza
- Switzerland (3):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Local Institution - 0189, Bellinzona
- Taiwan (6):
  - Local Institution - 0053, Kaohsiung City
  - Local Institution - 0050, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Local Institution - 0048, Taipei
  - Taipei Medical University Hospital, Taipei
  - Local Institution - 0160, Taipei
- Thailand (4):
  - Local Institution - 0265, Bangkok, Bangkok
  - Local Institution - 0272, Mueng, Changwat Khon Kaen
  - Local Institution - 0264, Bangkok
  - Local Institution - 0266, Songkhla
- United Kingdom (4):
  - Local Institution - 0110, Glasgow, Glasgow City
  - Local Institution - 0061, London, Kensington and Chelsea
  - Local Institution - 0140, London, London, City of
  - Local Institution - 0281, Sulton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07100080.html